CLINICAL TRIAL: NCT03067480
Title: Comparison of 3 Versus 6-Month Use of Professional Continuous Glucose Monitoring in the Treatment of Poorly Controlled, Non-Insulin Using T2DM Patients in a Primary Care Setting
Brief Title: Comparison of 3 Versus 6-Month Use of CGMS in Non-Insulin Using T2DM Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: East Tennessee State University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ETSU
Record Dates: First submitted 2017-02-24; First posted 2017-03-01 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 3-Month iPro2 Professional CGM (Experimental): Professional CGM measures interstitial glucose every 5 minutes via a glucose-oxidase-impregnated membrane during a 3 day period. The patient wearing professional CGM is blinded to the repeated measurements and the data is stored for retrospective analysis.
  Interventions: Device: iPro2 Professional CGM
- 6-Month iPro2 Professional CGM (Experimental): Professional CGM measures interstitial glucose every 5 minutes via a glucose-oxidase-impregnated membrane during a 3 day period. The patient wearing professional CGM is blinded to the repeated measurements and the data is stored for retrospective analysis.
  Interventions: Device: iPro2 Professional CGM

INTERVENTIONS:
Device: iPro2 Professional CGM — Professional CGM measures interstitial glucose every 5 minutes via a glucose-oxidase-impregnated membrane during a 3 day period. The patient wearing professional CGM is blinded to the repeated measurements and the data is stored for retrospective analysis.

SUMMARY:
To determine whether 3-month versus 6-month professional CGM utilization improves time spent in target range of 70-140mg/dl in patients with poorly controlled T2DM not treated with insulin.

DETAILED DESCRIPTION:
Patients not receiving any insulin treatment with an HbA1c ≥ 7.5% before their scheduled primary care appointment will be invited to participate in the study and wear professional CGM for at least 3 days at either 3 intervals (baseline, 3-month and 6-month) or 2 intervals (baseline and 6-month). After removal, the downloaded report will provide quantitative data to determine the percent of time spent in the target range. The 6-month data will be analyzed to determine if frequency of professional CGM wear positively affects time spent in target range.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older with a diagnosis of T2DM with a scheduled office visit with primary care provider within the next 4 weeks
2. Last 2 HbA1c values between 7.5 - 10% measured in the last 12 months
3. Treated with non-insulin therapies or therapeutic lifestyle changes
4. Never worn professional CGM or have not worn in last 12 months
5. Willing to perform requirements needed for professional CGM

Exclusion Criteria:

1. Current or previous treatment with any insulin within 3 months at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rick Hess, PharmD, Principal Investigator — East Tennessee State University
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3-Month iPro2 Professional CGM | 6-Month iPro2 Professional CGM
Started | 5 | 7
Completed | 2 | 2
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 2 | 4
Not completed — started insulin | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3-Month iPro2 Professional CGM | 6-Month iPro2 Professional CGM | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (4.8) | 54.0 (7.3) | 57.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
A1c [Mean (Standard Deviation); unit: percent] | 9.7 (1.6) | 9.6 (1.2) | 9.6 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Time Spent in Target Range
Description: Time sensor glucose is between 70-140mg/dl during a 72 hour collection period
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | 3-Month iPro2 Professional CGM | 6-Month iPro2 Professional CGM
Number analyzed (Participants) | 2 | 2
percentage | 38.5 (18.5) | 50 (40)

ADVERSE EVENTS:
Time Frame: 1 year
Description: no deaths reported
Arm/Group | 3-Month iPro2 Professional CGM | 6-Month iPro2 Professional CGM
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT03067480/Prot_SAP_001.pdf